CLINICAL TRIAL: NCT04265482
Title: GERO Cohort Protocol, Chile, 2017 - 2019: Community-based Cohort of Functional Decline in Subjective Cognitive Complaint Elderly
Brief Title: Community-based Cohort of Functional Decline in Subjective Cognitive Complaint Elderly
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Geroscience Center for Brain Health and Metabolism (Gero) (Other Government)
Responsible Party: Sponsor
Other Study IDs: FONDAP 15150012
Record Dates: First submitted 2020-02-03; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Subjective Cognitive Complaint; Activities Daily Living; Dementia; Alzheimer Disease; Neurodegenerative Diseases; Functionality; Gait Disorders, Neurologic; Geroscience
Keywords: Cognitive Ageing; Subjective Cognitive Complaint; Dementia; Alzheimer; Functional decline; Geroscience
MeSH Terms: conditions — Dementia; Alzheimer Disease; Neurodegenerative Diseases; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, buffy coat, plasma, serum, peripheral mononuclear cells, stool samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background With the global population aging and life expectancy increasing, dementia has turned a priority in the health care system. In Chile, dementia is one of the most important causes of disability in elderly, corresponding nearly to 40% of cases, and the most rapidly growing cause of death in the last twenty years. Cognitive complaints are considered a marker able to predict cognitive and functional decline, incident mild cognitive impairment (MCI), and incident dementia. The Gero cohort is the Chilean core clinical project of the Gerocenter on Brain Health and Metabolism (GERO), whose aim is to establish the capacity in Chile to foster cutting edge and multidisciplinary research on aging.

Objective This study has two main objectives. First, i) to analyze the rate of functional decline and progression to clinical dementia and their risks factors (biomedical, imaging, psychosocial, and clinical) in a community-dwelling elderly with subjective cognitive complaint, through a population-based study. Second, ii) to build the capacity to undertake clinical research on brain aging and dementia disorders and create Data-Bank and Bio-Banks with an appropriate infrastructure to further studies and facilitate access to the data and samples for research.

Methods The Gero cohort aims at recruiting 300 elderly subjects (>70 years) from the community of Santiago (Chile), following them up for at least 3 years. Eligible people are non-demented adults with subjective cognitive complaint, which are reported either by the participant, the proxy or both. Participants are identified through a household census. The protocol of evaluation is based on a multidimensional approach including socio-demographic, biomedical, psychosocial, neuropsychological, neuropsychiatric and motor assessments. Neuroimaging, blood and stool sample samples are also included. This multidimensional evaluation is carried out in a baseline assessment and 3 follow-ups assessment, at 18 and 36 months. In addition, in months 6, 24, and 30, a telephone interview is done in order to keep contact with the participants and to assess general well-being.

DETAILED DESCRIPTION:
Objectives of the Study:

The general objective of this study is to analyze the rate of functional decline (FD) and progression to clinical dementia and their risks factors (biomedical, imaging, psychosocial, and clinical) in a community-dwelling elderly with subjective cognitive complaint (SCC), through a population-based study. The specific objectives are to determinate (i) longitudinal evolution of biomarkers measured from blood, stool and structural and functional neuroimaging (MRI), (ii) evolution of the health-related quality of life; (iii) rate of cardiovascular events (stroke and coronary events), and (iv) mortality rates. The investigators also aim to build the capacity to undertake clinical research on brain aging and dementia disorders and create Data-Bank and Bio-Banks with an appropriate infrastructure to further studies and facilitate access to the data and samples for research.

The Gero cohort is the core clinical project of the GERO, supported by the Fund for Research Centers in Priority Areas Program (FONDAP) of the Chilean National Commission for Scientific and Technological Research (CONICYT). GERO is initially funded for 5 years, and its main aim is to establish a center for studying Brain Aging in Chile including basic and clinical research.

Methods/Design

Field work during the first contact

The recruitment process considers two steps. Firstly, a lay team contacts each home to determine the presence of eligible individuals. In positive cases, the person receives a second visit by a trained psychologist who proceeds to check the eligibility. In case of acceptance, the inclusion and exclusion criteria protocol are applied. If the subject fulfills the criteria, the psychologist schedule a medical interview. Following this evaluation, a neurologist decides if the subject fulfill the inclusion criteria of the cohort.

The fieldwork is preceded by an outreach campaign (flyers, local radio advertisements, and presentations to community-organized groups) raising awareness about the visit of interviewers and the relevance of participating in the study. Rates of contact and response are monitored permanently, and the procedures around the contact and first interview are checked in the field and also by telephone to a subsample of participants. Contact to homes is attempted up to three times on different days and hours before considering it frustrated. The fieldwork started in November 2017 and is expected to finish at the end of 2019.

The lay team and psychologists involved in the first contact and recruitment received specific training on their labour in the field. The lay team completed a whole week training, which included theoretical and practical elements. Psychologists received a twelve weeks length training, which covers several sessions of neuropsychological assessment, including performance psychology.

Sample size

The sample size had to satisfy two criteria, one concerned with the statistical power required to explore multiple associations with outcomes, and other related to the feasibility to perform a wide range of assessments to each participant assuming costs and logistics. Both criteria meant a trade-off between the tolerance to uncertainty around the parameters to be estimated and the number of assessments that would be investigated throughout the study. The final sample chosen was 300 participants. This number allows maintaining the integrity of the original protocol and permits to test associations equivalent to an odds ratio (OR) around 1.5 (Cohen's d equal to 0,22) in cases of exposition and probability of the outcome close to 50%, using a significance of 5%. It is expected to follow each participant between 2 and 3 years, accumulating roughly 750 person-years of follow up.

Follow-up and retention strategy

Socio-demographic, clinical, psychosocial, neuropsychological, neuropsychiatric, motor, neuroimaging, blood biomarkers, stool, and genetic samples will be performed as baseline evaluation and every 18 months, with the exception of genetic study that will be performed only at baseline and neuroimaging at baseline and the 36 month. Patients' health status, functionality, and involvement in the Gero cohort will be monitored every 6 months by a telephonic questionnaire.

To avoid a significant attrition of the sample a set following strategies have been considered: to recruit only people who have at least one person that can facilitate the contact with him or her, it means a person who can be contacted for asking about the location of the participant; telephone contact every six months; and domicile visit in case of absence of contact or attending to assessment appointments. Additionally, all transport costs of participants will be covered by the Gero cohort administration, as well as any food that is required during the days of assessment. Initially, the end of the follow up of the cohort is programmed for October 2022.

Assessments and measurements

The protocol considers an intensive and deep multidimensional study of factors related to the prognosis of FD and dementia development. The range of assessments includes: socio-demographic, psychosocial, neuropsychological, neuropsychiatric, motor, neuroimaging, blood biomarkers, genetic and stool samples to perform gut microbiome studies. Neuroimaging protocol will allow assessing brain atrophy, structural and functional connectivity and white matter lesions. Gero biological samples of whole blood, buffy coat, plasma, serum, and peripheral mononuclear cells are taken and processed according to the guidelines published in 2015. Samples are stored in our Gero biobank for long-term storage at -80 °C or in liquid nitrogen. Stool samples will be collected using standardized kits and DNA extracted using the protocol Q suggested by the international human microbiome standards (IHMS SOP 06 V1). Data are recorded in an ad-hoc platform developed by bioinformatics and bioengineers personal of Gero.

Data analysis plan

The Gero cohort offers a unique opportunity for multiple analyses to identify, correlate and analyze multidimensional factors related to FD and progression to dementia in elderlies with SCC.

In broad terms, a descriptive of baseline measurements (either outcomes or potential predictive factors) will be performed. The procedure will be repeated at each measurement time, every 18 months. Random effect models will be used for describing trajectories of participant subgroups and the whole cohort according to main variables, using Markov-Chain Montecarlo procedures.

The association between variables and outcomes will be explored broadly using different machine learning methods, such as elastic net procedure, random forest procedure, based-tree methods, and support vector machines. These procedures are suitable to lead with multi-collinearity and also high dimensional data (e.g. the number of predictive variables is larger than the number of participants in the cohort). Interpretation of causality will be conducted using standard random effect models and eventually structural equation modeling.

Missing data and loss of follow up of participants are common in observational studies, mainly in cohorts. Firstly, cases with missing data in any outcome will be explored and compared with cases without missing data describing any pattern. Secondly, two strategies will be followed to estimate results: (1) to analyze only cases with complete information (i.e. assuming that missing data is completely at random); and (2) imputing data according to multivariate imputation by chained equation techniques. The analysis will be performed using the statistical software R.

Coordination with local health services

The Gero cohort has been carefully design to avoid undermining the usual care of participants in their common health services facilities. Even more, a linkage between the health assessments provided by the cohort and the usual health care has been promoted.

In cases when the cohort's assessment detects a new health condition (diabetes, depression, hypertension, etc.), participants are derived to the primary healthcare centre of their territory. In case of detection of a significant neurological disorder (dementia syndrome, Parkinson, etc.) the participants are directly derived to specialized care according to their health district, communicating the decision to the primary health care.

Primary care health centres, specialized care polyclinics and the direction of the Health District involved have been informed about the study and jointly the protocol of derivation and communication were established.

Regulation of access to data/biospecimens

The access to data and biospecimens is regulated by the GERO directorate in accordance with the local Institutional Review Board authorization. A bilateral agreement must be signed before sharing of data. Access to the server will not be granted.

ELIGIBILITY:
Inclusion Criteria:

* 70 years old or older.
* Presence of a knowledgeable informant and/or presence of a contact that allows the follow up of the participant.
* Being affiliated to the public health insurance.
* Subjective cognitive complaint either self-reported or reported by a knowledgeable informant.
* Clinical Dementia Scale- frontotemporal lobar degeneration (CDR-FTLD) equal or inferior to 0.5.
* Signed informed consent

Exclusion Criteria:

* Report of medical diagnosis of dementia.
* Mini-mental State Examination (MMSE) < 21 and Pfeffer questionnaire >2.
* Institutionalization (for example, living in an elderly home or a skilled nursing facility)
* Illiteracy, meaning that is not able to count or to read.
* Visual and auditory acuity not adequate for neuropsychological testing.
* Important limitation of mobility incompatible with the availability to be independent in daily life activities or attending a clinical centre for further evaluation.
* Report of medical diagnosis of Parkinson's disease.
* Report of medical diagnosis of one or more of the following conditions causing severe impairment in functionality: any psychiatric or neurological disorders, brain tumor, subdural haematoma, progressive supranuclear palsy, or history of head trauma.
* Report of medical diagnosis of stroke occurred in the last three months.
* Presence of a fatal disease (less than one year of survival)

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The cohort recruits the potential participants from the general population, using a door-to-door strategy. The sample framework corresponds to the territories assigned to three primary healthcare centres selected by convenience according to their socioeconomic heterogeneity, which belong to three different districts in Santiago (Chile): Macul, Peñalolen and La Reina. The sample considered a two-stage selection process. The first stage included a sample of quadrants within each territory, where the contact to all houses was attempted. The second stage proceeded when in a home was found more than one potential eligible participant, choosing one randomly. Territories encompassed a population between 14,937 and 39,458 people. of which between 4.6% and 8.0% is expected to be older than 70.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-09-25 (Actual); Primary Completion 2020-09-25 (Estimated); Study Completion 2023-09-25 (Estimated)

PRIMARY OUTCOMES:
Rate of functional decline and progression to clinical dementia | Changes from baseline at 18 and 36 months.
  The protocol considers an intensive and deep multidimensional study of factors related to the prognosis of functional decline and dementia development. The range of assessments includes: sociodemographic, psychosocial, neuropsychological, neuropsychiatric, motor, neuroimaging, blood biomarkers, genetic and stool samples to perform gut microbiome studies.

SECONDARY OUTCOMES:
Longitudinal evolution of biomarkers and functional neuroimaging (fMRI) | Changes from baseline at 18 and 36 months.
  Gero biological samples of whole blood, buffy coat, plasma, serum, and peripheral mononuclear cells are taken and processed according to the guidelines published in 2015. Samples are, stored in our Gero biobank for long-term storage at -80 °C or in liquid nitrogen. Stool samples will be collected using standardized kits and DNA extracted using the protocol Q suggested by the international human microbiome standards (IHMS SOP 06 V1). Neuroimaging protocol will allow assessing brain atrophy, structural and functional connectivity and white matter lesions.
Evolution of the health-related quality of life: EQ3D | Changes from baseline at 18 and 36 months.
  Health related quality of life will be assessed using the EQ3D and monitored by a period telephone contact. EQ3D is a standardized instrument for measuring generic health status, where 0% is the worst possible health self-perception and 100% is the best health self-perception.
Rate of cardiovascular events | Changes from baseline at 18 and 36 months.
Mortality rates | Changes from baseline at 18 and 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Slachevsky, MD, Principal Investigator — Geroscience Center for Brain health and Metabolism
Locations (1):
- Universidad de Chile, Santiago, Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pievani M, Filippini N, van den Heuvel MP, Cappa SF, Frisoni GB. Brain connectivity in neurodegenerative diseases--from phenotype to proteinopathy. Nat Rev Neurol. 2014 Nov;10(11):620-33. doi: 10.1038/nrneurol.2014.178. Epub 2014 Oct 7. PMID 25287597
- [Background] Ferrarini L, van Lew B, Reiber JH, Gandin C, Galluzzo L, Scafato E, Frisoni GB, Milles J, Pievani M; IPREA Working Group (Italian PRoject on Epidemiology of Alzheimer's disease). Hippocampal atrophy in people with memory deficits: results from the population-based IPREA study. Int Psychogeriatr. 2014 Jul;26(7):1067-81. doi: 10.1017/S1041610213002627. Epub 2014 Feb 13. PMID 24524645
- [Background] O'Bryant SE, Gupta V, Henriksen K, Edwards M, Jeromin A, Lista S, Bazenet C, Soares H, Lovestone S, Hampel H, Montine T, Blennow K, Foroud T, Carrillo M, Graff-Radford N, Laske C, Breteler M, Shaw L, Trojanowski JQ, Schupf N, Rissman RA, Fagan AM, Oberoi P, Umek R, Weiner MW, Grammas P, Posner H, Martins R; STAR-B and BBBIG working groups. Guidelines for the standardization of preanalytic variables for blood-based biomarker studies in Alzheimer's disease research. Alzheimers Dement. 2015 May;11(5):549-60. doi: 10.1016/j.jalz.2014.08.099. Epub 2014 Oct 1. PMID 25282381
- [Background] Browne, W.J., MCMC Estimation in MLwiN (Version 2.13) Centre for Multilevel Modelling. 2015, Bristol, UK: Centre for Multilevel Modelling, University of Bristol.
- [Background] Christensen, R., et al., Bayesian Ideas and Data Analysis: An Introduction for Scientists and Statisticians. . 2010, U.S.A: CRC Press
- [Background] James, G., et al., An Introduction to Statistical Learning with Applications in R. . Springer Texts in Statistics. 2017: Springer.
- [Background] Hoyle, R.H., Handbook of Structural Equation Modeling. . 2012: The Guilford Press.
- [Background] Steyerberg, E., Clinical Prediction Model: Ch. 8: Case Study on Dealing with Missing Data. Statistics for Biology and Health, 2009: p. 139 - 158.
- [Background] Steyerberg, E., Clinical Prediction Models: Ch. 7: A Practical Approach to Development, Validation, and Updating. Statistics for Biology and Health, 2009: p. 115 - 137.
- [Derived] Slachevsky A, Zitko P, Martinez-Pernia D, Forno G, Court FA, Lillo P, Villagra R, Duran-Aniotz C, Parrao T, Assar R, Orellana P, Toledo C, Rivera R, Ibanez A, Parra MA, Gonzalez-Billault C, Amieva H, Thumala D. GERO Cohort Protocol, Chile, 2017-2022: Community-based Cohort of Functional Decline in Subjective Cognitive Complaint elderly. BMC Geriatr. 2020 Nov 25;20(1):505. doi: 10.1186/s12877-020-01866-4. PMID 33238908